CLINICAL TRIAL: NCT06304545
Title: Long-course Concurrent Chemoradiotherapy Combined With Camrelizumab in the Neoadjuvant Treatment of Locally Advanced/Low Anus-preserving Rectal Cancer: a Phase II Single-arm Study.
Brief Title: Treatment of Rectal Cancer With Long-term Concurrent Chemoradiotherapy Combined With Camrelizumab
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Chunbo Zhao, Principal Investigator, Harbin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-HLJ-081
Record Dates: First submitted 2024-03-01; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Rectal Cancer
Keywords: Camrelizumab; Long-term concurrent chemoradiotherapy; Neoadjuvant treatment; Locally advanced/low cancer requiring anus preservation
MeSH Terms: conditions — Rectal Neoplasms | interventions — camrelizumab; Drug Therapy; Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemoradiotherapy combined with immunotherapy for early rectal cancer. (Experimental): Radiotherapy and Chemotherapy combined with Camrelizumab
  Interventions: Drug: Camrelizumab; Drug: Chemotherapy; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab IV 200mg
  Other Names: SHR-1210
Drug: Chemotherapy — Capecitabine PO oxaliplatin IV
  Other Names: Capecitabine or combined oxaliplatin
Radiation: Radiotherapy — Radiotherapy 50Gy /45Gy /25 fractions
  Other Names: Long-term concurrent chemoradiotherapy

SUMMARY:
This is a single-arm, phase II clinical study aim to evaluate the efficacy and safety of long-term concurrent chemoradiotherapy combined with camrelizumab as a neoadjuvant therapy in the treatment of locally advanced/low rectal cancer requiring anus preservation.

DETAILED DESCRIPTION:
This study plans to recruit 48 patients with locally advanced/low anal preservation requiring rectal cancer. The study aims to observe and evaluate the efficacy and safety of long-term concurrent chemoradiotherapy combined with camrelizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 75 years old, male or female,
2. Histologically or cytologically confirmed rectal cancer with measurable tumour lesions (Spiral CT or MR scans ≥ 10 mm, meeting RECIST 1.1 criteria),
3. Clinical stage: Rectal cancer cT3-4N0M0 or cT1-4N+M0 and low rectal cancer with need for anal preservation (<5 cm from anal verge; T2N0M0),
4. Expected survival > 3 months,
5. ECOG PS score: 0-1,
6. No peritoneal metastasis or other distant metastasis; Note: the presence of distant metastasis should be confirmed by CT or MR scan. If bone metastasis is suspected, a bone scan should be performed. If peritoneal metastasis is suspected, PET-CT should be performed or laparoscopy should be performed. If brain metastases are suspected, CT or MR should be performed,
7. No previous radiotherapy or immune checkpoint inhibitor treatment for rectal cancer,
8. Function of vital organs in accordance with the following requirements (excluding the use of any blood components and cell growth factors during screening):

1)Absolute neutrophil count ≥ 1.5 x 10^9/L; platelets ≥ 80 x 10^9/L; hemoglobin ≥ 8.5 g/dL, 2)Thyroid-stimulating hormone (TSH) ≤1 times ULN (if abnormal, T3 and T4 levels should be examined at the same time; if T3 and T4 levels are normal, they can be enrolled), 3)Bilirubin ≤1.5 times ULN; ALT and AST ≤2.5 times ULN, 4) Serum creatinine ≤1.5 times ULN, 9. Women of childbearing potential must undergo a negative pregnancy test (βHCG) prior to initiation of treatment, and women of childbearing potential and men who are sexually active with women of childbearing potential must agree to use effective contraception uninterruptedly for the duration of the treatment period and for 6 months after the administration of the last therapeutic dose, 10. Subjects voluntarily enrolled in the study and signed an informed consent form.

Exclusion Criteria:

1. Previous pelvic or abdominal radiotherapy,
2. Tumours that are expected to be unresectable after neoadjuvant therapy,
3. Pregnant or lactating women, or those of childbearing potential who refuse to use contraception,
4. History of other malignancies within the past 5 years, except adequately treated carcinoma in situ of the cervix or squamous carcinoma of the skin, or basal cell carcinoma of the skin that has been substantially controlled,
5. Ineffectively controlled, symptomatic brain metastases or a history of psychosis that cannot be easily controlled or severe intellectual or cognitive dysfunction,
6. Pulmonary fibrosis, interstitial pneumonitis, pneumoconiosis, radiation pneumonitis, drug-associated pneumonitis and severely impaired lung function,
7. Subjects with active, known or suspected autoimmune disease, hypothyroidism requiring only hormone replacement therapy, skin disorders that do not require systemic therapy (e.g., vitiligo, psoriasis, or alopecia areata) may be eligible for enrolment,
8. Congestive heart failure, difficult-to-control cardiac arrhythmia, myocardial infarction within 6 months, unstable angina, stroke or transient is chaemic attack, severe hypertension difficult to control with medication, or other patients who cannot tolerate the procedure,
9. Severe active infections requiring intravenous antibiotic treatment occurring during the screening period,
10. Allergy to the test drug,
11. Have received or will receive a live vaccine within 30 days prior to camrelizumab administration,
12. Known history of HIV infection or active hepatitis B or C,
13. Patients who are unable to comply with the trial protocol or are unable to cooperate with follow-up visits,
14. Those who in the opinion of the investigator are not suitable for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2026-08-16 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response rate | up to 24 months
  After neoadjuvant therapy and surgery, postoperative specimens showed no residual surviving tumor cells in the tumor bed (%RVT=0).

SECONDARY OUTCOMES:
Objective Response Rate | up to 24 months
  Determined using RECIST v1.1 criteria, defined as best overall response (CR or PR) across all assessment time points during the period from enrolment to termination of trial treatment.
Disease Control Rate | up to 24 months
  Determined using RECIST v1.1 criteria.
Anal preservation rate | up to 24 months
  Proportion of patients with low rectal cancer who retain their anus after surgery.
Disease-free Survival | up to 24 months
  The time from surgical resection to the first tumor recurrence and metastasis, or the patient's death due to any reason.
Overall Survival | up to 36 months
  Defined as the time from randomizstion to death from any cause.
AEs | up to 24 months
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0.
3-years Overall Survival rate | up to 36 months
  Proportion of death from randomization to 3 years of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Chunbo Zhao, MD, Principal Investigator — Harbin Medical University Cancer Hosptital

IPD SHARING:
Plan to Share IPD: No